CLINICAL TRIAL: NCT04225832
Title: A Cognitive Behavioral Therapy Group Intervention to Increase HIV Testing and PrEP Use Among Latinx Sexual Minority Men
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Government executive order
Sponsor: RAND (Other)
Collaborators: Bienestar Human Services, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01MH121256 (NIH)
Record Dates: First submitted 2020-01-07; First posted 2020-01-13 (Actual); Results first posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2023-11

CONDITIONS: HIV
Keywords: Latino/Hispanic/Latinx; men who have sex with men
MeSH Terms: conditions — Homosexuality

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor does not randomize participant until after the baseline assessment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT Coping Intervention (Experimental): The intervention is an 8-session cognitive behavior therapy (CBT) group intervention that aims to improve HIV outcomes by increasing adaptive, effective coping responses to stigma from intersectional identities related to ethnicity, immigration status, sexual minority identity, HIV status, and PrEP among Latinx sexual minority men (SMM). The intervention sessions will address topics such as: understanding and coping with intersectional stigma, multiple identities (e.g., race/ethnicity, sexual orientation), medical mistrust, social support, and structural stigma. Intervention groups will be led by a trained facilitator (with expertise in group therapy with Latinx SMM) and a trained peer co-facilitator matched in identities with participants (Latinx SMM).
  Interventions: Behavioral: CBT Coping Intervention
- Control (No Intervention): Participants who are randomized to the control condition will be referred to the standard of care program at Bienestar, which includes an ongoing weekly open wellness-oriented support group available to all clients.

INTERVENTIONS:
Behavioral: CBT Coping Intervention — A cognitive behavior therapy group intervention for HIV-negative Latinx sexual minority men aimed at increasing HIV testing and prevention strategies.
  Arms: CBT Coping Intervention

SUMMARY:
This study consists of a randomized controlled trial (RCT) of a multi-session cognitive behavior therapy (CBT) group intervention that aims to improve HIV outcomes by increasing adaptive, effective coping responses to stigma from intersectional identities related to ethnicity, immigration status, sexual minority identity, HIV status, and PrEP use among Latinx sexual minority men (SMM).

DETAILED DESCRIPTION:
This study consists of a randomized controlled trial (RCT) of a multi-session cognitive behavior therapy (CBT) group intervention that aims to improve HIV outcomes by increasing adaptive, effective coping responses to stigma from intersectional identities related to ethnicity, immigration status, sexual minority identity, HIV status, and PrEP use among Latinx sexual minority men (SMM). We will test intervention effects on regular HIV testing and use of prevention strategies. The intervention was developed in partnership with community stakeholders at Bienestar Human Services, Inc., a Latinx-focused organization in Los Angeles County (LAC), CA. The intervention is flexible for use in community-based organizations, such as in ongoing support groups.

The Specific Aims are:

Aim 1. To conduct a randomized controlled trial of a culturally congruent cognitive behavior therapy group intervention for immigrant Latinx sexual minority men, to test intervention effects on regular HIV testing and PrEP uptake.

Aim 2. To examine mechanisms of intervention effects on regular HIV testing and PrEP uptake, including more effective coping (e.g., reduced internalized stigma).

Aim 3. To conduct a cost-effectiveness analysis of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years-old
* biologically male at birth
* identify as male
* identify as Latino
* is an immigrant
* report having sex with men in the past 12 months
* report HIV-negative or unknown serostatus
* anticipate being available for the next 12 months to attend study visits
* able to interact and communicate in spoken Spanish or English.

Exclusion Criteria:

* HIV-positive
* cisgender women
* transgender women

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — * biologically male at birth
  * identify as male
Enrollment: 289 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2024-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Bogart, PhD, Principal Investigator — RAND
Locations (1):
- Bienestar Human Services, Inc, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited across Southern California using: in-person in-reach at the partner organization; in-person outreach at relevant events and businesses; passive recruitment via hard copy fliers left at the partner community-based organization and other relevant local organizations; social media recruitment via paid advertisements, video posts, and direct messaging. Participants also were offered $10 per referral, for up to three referrals.
Pre-assignment Details: Of 607 screened, 455 met inclusion criteria, of whom 289 were randomized.
Groups:
- Control: Participants who are randomized to the control condition will receive standard of care
Period: Overall Study
Arm/Group | CBT Coping Intervention | Control
Started | 145 | 144
Completed | 103 | 136
Not Completed | 42 | 8
Not completed — No longer eligible (e.g., seroconversion) | 6 | 3
Not completed — Unable to recontact or too busy/not recontacted or unknown reason | 36 | 5

BASELINE CHARACTERISTICS:
Population: 9 withdrawn (3 control, 6 intervention); 41 no follow-up data (5 control, 36 intervention) Analysis sample = 136 control, 103 intervention
Groups:
- Total: Total of all reporting groups
Arm/Group | CBT Coping Intervention | Control | Total
Number analyzed (Participants) | 145 | 144 | 289
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.3 (9.8) | 37.5 (10.0) | 37.9 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 145 | 144 | 289
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 145 | 144 | 289
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 145 | 142 | 287
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 145 | 144 | 289
HIV testing in past 12 months [Count of Participants; unit: Participants] — Population: Data missing for n=7 participants who did not answer whether they had ever had an HIV test or who did not provide the date of their last test
  Participants
    number analyzed (Participants) | 141 | 141 | 282
    (all) | 86 | 81 | 167
Current PrEP use [Count of Participants; unit: Participants] | 40 | 43 | 83
Brief COPE: Social support-seeking [Mean (Standard Deviation); unit: scores on a scale] — Participants completed the Brief COPE, a general measure of coping strategies. Items have the instruction "indicate the extent you do what the item says when you are faced with discrimination," and response options 1 = "I haven't been doing this at all," 2 = "I've been doing this a little bit," 3 = "I've been doing this a medium amount" and 4 = "I've been doing this a lot." This scale (identified by EFA) is the mean of 4 items such as "I get emotional support from others". Cronbach's alpha = .79.
  Higher values indicate more use of these coping strategies. Population: Coping missing for n=2 who did not respond to any of the 4 survey items in the scale
  scores on a scale
    number analyzed (Participants) | 145 | 142 | 287
    (all) | 2.12 (.86) | 2.28 (.90) | 2.20 (0.88)

OUTCOME MEASURES:

1. Primary Outcome: HIV Test at Least Annually
Description: Participants report being tested for HIV at least once in the 12 months after baseline
Time Frame: from baseline to 12-months
Measure: Count of Participants; unit: Participants
Arm/Group | CBT Coping Intervention | Control
Number analyzed (Participants) | 103 | 136
Participants | 96 | 114
Statistical Analysis 1: Comparison: CBT Coping Intervention vs Control; Test type: Superiority; p = .049, Regression, Logistic — a-priori threshold was p<.05 for two-sided p-value Regression employed nonresponse weights to account for any bias associated with completing any follow-up survey; Regression results control for immigration status and length of time in U.S; Odds Ratio (OR) = 2.51, 95% CI 2-sided [1.01 to 6.26] — Odds ratio is for indicator of intervention arm; Regression results control for immigration status and length of time in U.S

2. Primary Outcome: Took PrEP in the Past 12 Months
Description: Participants report taking PrEP at any follow-up time-point (within the 12-month follow-up time period)
Time Frame: from baseline to 12-months
Population: Of the N=289 described in Baseline Characteristics, N=50 did not complete any follow up assessments. Outcome measures are assessed for the remaining N=239
Measure: Count of Participants; unit: Participants
Arm/Group | CBT Coping Intervention | Control
Number analyzed (Participants) | 103 | 136
Participants | 56 | 71
Statistical Analysis 1: Comparison: CBT Coping Intervention vs Control; Test type: Superiority; p = .83, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Regression results control for immigration status and length of time in U.S; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.62 to 1.81] — Odds ratio is for indicator of intervention arm

3. Secondary Outcome: Level of Adaptive Coping
Description: Participants completed the Brief COPE, a general measure of coping strategies. Items have the instruction "indicate the extent you do what the item says when you are faced with discrimination," and response options 1 = "I haven't been doing this at all," 2 = "I've been doing this a little bit," 3 = "I've been doing this a medium amount" and 4 = "I've been doing this a lot." This scale (identified by EFA) is the mean of 4 items such as "I get emotional support from others".
  Higher values indicate more use of these coping strategies.
Time Frame: measured at 4-months, 8-months, and 12-months post baseline
Population: Of the N=289 described in Baseline Characteristics, N=50 did not complete any follow up assessments. An additional N=2 control participants did not respond to any of the 4 items in the scale, leaving N=237 for analysis
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | CBT Coping Intervention | Control
Number analyzed (Participants) | 103 | 134
scores on a scale
  4-month assessment: number analyzed (Participants) | 95 | 128
  4-month assessment | 2.14 (0.96) | 2.05 (0.89)
  8-month assessment: number analyzed (Participants) | 83 | 112
  8-month assessment | 2.04 (0.84) | 2.02 (0.91)
  12-month assessment: number analyzed (Participants) | 101 | 116
  12-month assessment | 2.02 (0.92) | 1.96 (0.92)
Statistical Analysis 1: Comparison: CBT Coping Intervention vs Control; Unlike the "observed at any FU" primary outcomes which have a single value for each participant, for this outcome we employed a repeated measures style structure with one record for each of up to 3 FU observations. A sandwich estimator (SAS Proc Surveyreg) was employed to account for clustering of observations within participant; Test type: Superiority; p = .14, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Regression results control for immigration status, length of time in U.S., and baseline value of the outcome; Slope = 0.14, Standard Error of Mean .09 — Slope is adjusted regression coefficient for indicator of intervention arm

ADVERSE EVENTS:
Time Frame: 3 years, 9 months
Arm/Group | CBT Coping Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/145 | 0/144
Serious Adverse Events (participants affected / at risk) | 21/145 | 3/144
Other Adverse Events (participants affected / at risk) | 0/145 | 0/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CBT Coping Intervention (N=145) | Control (N=144)
Potential confidentiality breach (Social circumstances) | 14 (14) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 5 (5) | 1 (1)
social threat/violence (Social circumstances) | 1 (1) | 1 (1)
Surgery due to pre-existing condition (Surgical and medical procedures) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Objective HIV testing dates and PrEP prescription data were collected (e.g., from medical records), but the US federal government (NIH) terminated the grant prematurely on March 20, 2025 before these data could be processed. These data were not fully cleaned or tabulated, and thus were not analyzed as an outcome and cannot be entered at baseline: The number of records is unknown and therefore not reported here. Thus, the primary outcomes are reported based on self-reported survey responses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-06): https://cdn.clinicaltrials.gov/large-docs/32/NCT04225832/Prot_SAP_000.pdf